CLINICAL TRIAL: NCT03347110
Title: A Multicenter, Open-Label, Follow-Up Study to Evaluate the Long-Term Safety and Efficacy of Bimekizumab in Subjects With Psoriatic Arthritis
Brief Title: A Study to Evaluate the Long-Term Safety and Efficacy of Bimekizumab in Subjects With Psoriatic Arthritis
Acronym: BE ACTIVE 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma SRL (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA0009; 2017-001003-74 (EudraCT Number)
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Results first posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Psoriatic Arthritis
Keywords: Bimekizumab; Psoriatic Arthritis; PsA
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — bimekizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bimekizumab (Experimental): Subjects will receive bimekizumab up to 2 years.
  Interventions: Drug: Bimekizumab

INTERVENTIONS:
Drug: Bimekizumab — Bimekizumab at a prespecified dose.
  Other Names: UCB4940

SUMMARY:
This is a study to assess the long-term safety and tolerability of bimekizumab in subjects with psoriatic arthritis

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the Investigator, the subject is expected to benefit from participation in an Open Label Extension (OLE) study
* Subject completed PA0008 without meeting any withdrawal criteria
* Female subjects must be postmenopausal, permanently sterilized or, if of childbearing potential, must be willing to use a highly effective method of contraception
* Male subjects with a partner of childbearing potential must be willing to use a condom when sexually active

Exclusion Criteria:

* Female subjects who plan to become pregnant during the study or within 20 weeks following the last dose of IMP. Male subjects who are planning a partner pregnancy during the study or within 20 weeks following the last dose
* Subjects with any current sign or symptom that may indicate a medically significant active infection (except for the common cold) or has had an infection requiring systemic antibiotics within 2 weeks of study entry
* Subjects who meet any withdrawal criteria in PA0008. For any subject with an ongoing Serious Adverse Event, or a history of serious infections (including hospitalizations) in the lead-in study, the Medical Monitor must be consulted prior to the subject's entry into PA0009

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 8445992273 (UCB)
Locations (37):
- United States (11):
  - Pa0009 025, Lexington, Kentucky
  - Pa0009 003, Hagerstown, Maryland
  - Pa0009 011, Lansing, Michigan
  - Pa0009 028, Rochester, New York
  - Pa0009 014, Portland, Oregon
  - Pa0009 001, Duncansville, Pennsylvania
  - Pa0009 012, Johnston, Rhode Island
  - Pa0009 004, Charleston, South Carolina
  - Pa0009 010, Jackson, Tennessee
  - Pa0009 006, Dallas, Texas
  - Pa0009 013, Mesquite, Texas
- Czechia (6):
  - Pa0009 205, Brno
  - Pa0009 207, Olomouc
  - Pa0009 201, Prague
  - Pa0009 202, Prague
  - Pa0009 210, Prague
  - Pa0009 203, Zlín
- Germany (4):
  - Pa0009 302, Cologne
  - Pa0009 309, Erlangen
  - Pa0009 304, Hamburg
  - Pa0009 301, Ratingen
- Hungary (2):
  - Pa0009 403, Budapest
  - Pa0009 401, Veszprém
- Poland (9):
  - Pa0009 452, Bialystok
  - Pa0009 453, Elblag
  - Pa0009 456, Elblag
  - Pa0009 455, Krakow
  - Pa0009 451, Poznan
  - Pa0009 450, Torun
  - Pa0009 454, Warsaw
  - Pa0009 459, Warsaw
  - Pa0009 465, Wroclaw
- Russia (5):
  - Pa0009 604, Moscow
  - Pa0009 605, Moscow
  - Pa0009 607, Moscow
  - Pa0009 606, Saint Petersburg
  - Pa0009 608, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mease PJ, Asahina A, Gladman DD, Tanaka Y, Tillett W, Ink B, Assudani D, de la Loge C, Coarse J, Eells J, Gossec L. Effect of bimekizumab on symptoms and impact of disease in patients with psoriatic arthritis over 3 years: results from BE ACTIVE. Rheumatology (Oxford). 2023 Feb 1;62(2):617-628. doi: 10.1093/rheumatology/keac353. PMID 35789257
- [Derived] Mease PJ, Gensler LS, Orbai AM, Warren RB, Bajracharya R, Ink B, Marten A, Massow U, Shende V, Manente M, Peterson L, White K, Landewe R, Poddubnyy D. Long-term safety of bimekizumab in adult patients with axial spondyloarthritis or psoriatic arthritis: pooled results from integrated phase IIb/III clinical studies. RMD Open. 2025 Apr 6;11(2):e005026. doi: 10.1136/rmdopen-2024-005026. PMID 40194794
- [Derived] Coates LC, McInnes IB, Merola JF, Warren RB, Kavanaugh A, Gottlieb AB, Gossec L, Assudani D, Bajracharya R, Coarse J, Ink B, Ritchlin CT. Safety and Efficacy of Bimekizumab in Patients With Active Psoriatic Arthritis: Three-Year Results From a Phase IIb Randomized Controlled Trial and Its Open-Label Extension Study. Arthritis Rheumatol. 2022 Dec;74(12):1959-1970. doi: 10.1002/art.42280. Epub 2022 Nov 18. PMID 35829656

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in November 2017 and concluded in October 2020.
Pre-assignment Details: Participant Flow refers to the Safety Set. Participants who completed the study PA0008 (NCT02969525) were eligible to enroll in study PA0009. A total of 184 participants from PA0008 signed the Informed Consent Form and were enrolled in PA0009 study. Among 184 participants, 1 participant did not receive treatment and was not included in analysis.
Groups:
- Bimekizumab 160 mg: Participants received bimekizumab (BKZ) 160 milligrams (mg) as a subcutaneous (sc) injection every 4 weeks (Q4W) for up to 100 weeks.
Period: Overall Study
Arm/Group | Bimekizumab 160 mg
Started | 183
Completed | 161
Not Completed | 22
Not completed — Other (Participant is incarcerated) | 1
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 1
Not completed — Lack of Efficacy | 2
Not completed — Adverse Event, non-fatal | 9

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to SS which consisted of all study participants who had given informed consent for PA0009 and had received at least one dose of study medication in PA0009.
Groups:
- Bimekizumab 160 mg (SS): Participants received BKZ 160 mg as a sc injection Q4W for up to 100 weeks. Participants formed the Safety Set (SS) which consisted of all study participants who had given informed consent for PA0009 and had received at least one dose of study medication in PA0009.
Arm/Group | Bimekizumab 160 mg (SS)
Number analyzed (Participants) | 183
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 165
  >=65 years | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.0 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87
  Male | 96
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 4
  White | 179

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) During the Study
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. TEAEs were defined as events with onset date on or after the start date of study medication in PA0009.
Time Frame: From Entry Visit of PA0009 until Safety Follow-Up Visit (up to Week 120)
Population: The Safety Set (SS) consisted of all study participants who had given informed consent for PA0009 and had received at least one dose of study medication in PA0009.
Measure: Number; unit: percentage of participants
Groups:
- Bimekizumab 160 mg (SS): Participants received BKZ 160 mg as a sc injection Q4W for up to 100 weeks. Participants formed the SS which consisted of all study participants who had given informed consent for PA0009 and had received at least one dose of study medication in PA0009.
Arm/Group | Bimekizumab 160 mg (SS)
Number analyzed (Participants) | 183
percentage of participants | 80.9

2. Primary Outcome: Percentage of Participants With Treatment-emergent Serious Adverse Events (SAEs) During the Study
Description: A serious adverse event (SAE) was any untoward medical occurrence that at any dose resulted in death, life-threatening, significant or persistent disability/incapacity, congenital anomaly/birth defect, important medical event, initial inpatient hospitalization or prolongation of hospitalization.
Time Frame: From Entry Visit of PA0009 until Safety Follow-Up Visit (up to Week 120)
Population: The SS consisted of all study participants who had given informed consent for PA0009 and had received at least one dose of study medication in PA0009.
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 160 mg (SS)
Number analyzed (Participants) | 183
percentage of participants | 7.7

3. Secondary Outcome: Percentage of Participants Who Withdrew Due to Treatment-emergent Adverse Event (TEAE) During the Study
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Time Frame: From Entry Visit of PA0009 until Safety Follow-Up Visit (up to Week 120)
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 160 mg (SS)
Number analyzed (Participants) | 183
percentage of participants | 4.9

4. Secondary Outcome: Percentage of Participants With American College of Rheumatology 20% Improvement (ACR20) Response at Week 48 Calculated Relative to Baseline of PA0008
Description: The ACR20 response rate was based on 20% or greater improvement relative to Baseline of PA0008 in the following measures: Tender Joint Count (TJC) based on 78 joints, Swollen Joint Count (SJC) based on 76 joints; 3 of the 5 remaining core set measures: Disease activity as assessed by Patient's Global Assessment of Disease Activity (PGADA), Disease activity as assessed by Physician's Global Assessment of Disease Activity (PhGADA), Pain as assessed by Patient's Assessment of Arthritis Pain (PtAAP), Physical function as assessed by Health Assessment Questionnaire - Disability Index (HAQ-DI), Acute phase response as assessed by high sensitivity C-reactive protein (hs CRP). Participants for whom ACR could not be derived due to missing data were counted as non-responders as per NRI analysis.
Time Frame: Baseline of PA0008, Week 48
Population: The Full Analysis Set (FAS) consisted of all enrolled participants who received at least 1 dose of study medication in PA0009 and had a valid measurement for at least 1 efficacy variable after PA0009 entry visit.
Measure: Number; unit: percentage of participants
Groups:
- Bimekizumab 160 mg (FAS): Participants received BKZ 160 mg as a sc injection Q4W for up to 100 weeks. Participants formed the Full Analysis Set (FAS) which consisted of all enrolled participants who received at least 1 dose of study medication in PA0009 and had a valid measurement for at least 1 efficacy variable after PA0009 entry visit.
Arm/Group | Bimekizumab 160 mg (FAS)
Number analyzed (Participants) | 181
percentage of participants | 79.0

5. Secondary Outcome: Percentage of Participants With American College of Rheumatology 50% Improvement (ACR50) Response at Week 48 Calculated Relative to Baseline of PA0008
Description: The ACR50 response rate was based on 50% or greater improvement relative to Baseline of PA0008 in the following measures: TJC based on 78 joints, SJC based on 76 joints; 3 of the 5 remaining core set measures: Disease activity as assessed by PGADA, Disease activity as assessed by PhGADA, Pain as assessed by PtAAP, Physical function as assessed by HAQ-DI, Acute phase response as assessed by hs CRP. Participants for whom ACR could not be derived due to missing data were counted as non-responders as per NRI analysis.
Time Frame: Baseline of PA0008, Week 48
Population: The FAS consisted of all enrolled participants who received at least 1 dose of study medication in PA0009 and had a valid measurement for at least 1 efficacy variable after PA0009 entry visit.
Measure: Number; unit: percentage of participants
Groups:
- Bimekizumab 160 mg (FAS): Participants received BKZ 160 mg as a sc injection Q4W for up to 100 weeks. Participants formed the FAS which consisted of all enrolled participants who received at least 1 dose of study medication in PA0009 and had a valid measurement for at least 1 efficacy variable after PA0009 entry visit.
Arm/Group | Bimekizumab 160 mg (FAS)
Number analyzed (Participants) | 181
percentage of participants | 64.6

6. Secondary Outcome: Percentage of Participants With American College of Rheumatology 70% Improvement (ACR70) Response at Week 48 Calculated Relative to Baseline of PA0008
Description: The ACR70 response rate was based on 70% or greater improvement relative to Baseline of PA0008 in the following measures: TJC based on 78 joints, SJC based on 76 joints; 3 of the 5 remaining core set measures: Disease activity as assessed by PGADA, Disease activity as assessed by PhGADA, Pain as assessed by PtAAP, Physical function as assessed by HAQ-DI, Acute phase response as assessed by hs CRP. Participants for whom ACR could not be derived due to missing data were counted as non-responders as per NRI analysis.
Time Frame: Baseline of PA0008, Week 48
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 160 mg (FAS)
Number analyzed (Participants) | 181
percentage of participants | 47.5

7. Secondary Outcome: Change From Baseline of PA0008 in Maastricht Ankylosing Spondylitis Enthesitis Index (MASES) at Week 48 Calculated Relative to Baseline of PA0008
Description: The MASES is an index that measures the severity (ie, intensity and extent) of enthesitis through the assessment of 13 entheses (bilateral costochondral 1, costochondral 7, anterior superior iliac spine, posterior iliac spine, iliac crest and proximal insertion of the Achilles tendon sites, and the fifth lumbar vertebral body spinous process). Each item was scored as 0 = not tender or 1 = tender and then were summed for a possible score of 0 to 13, with higher scores indicating worse enthesitis. If 7 or more items were available, MASES was calculated by dividing the summed score with the number of assessments and multiplying the result by 13. If less than 7 items were available, MASES was treated as missing.
Time Frame: Baseline of PA0008, Week 48
Population: Subset of study participants in the FAS with Enthesitis at PA0008 Baseline (MASES>0).
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Bimekizumab 160 mg (FAS)
Number analyzed (Participants) | 95
score on a scale | -2.99 (0.33)

8. Secondary Outcome: Change From Baseline of PA0008 in the Leeds Dactylitis Index (LDI) at Week 48 Calculated Relative to Baseline of PA0008
Description: Presence of dactylitis was assessed using the LDI basic which evaluated for a greater than or equal to (>=) 10% difference in the circumference of the digit compared to the opposite digit and was then multiplied by the tenderness score, using a simple grading system (0=absent, 1=present). The results from each digit with dactylitis were summed to produce a final score. For the final score, the minimum value for LDI is zero and there is no maximum value. A low score indicates less dactylitis symptoms. A score of zero is considered dactylitis free. Observed values have been reported in this outcome measure.
Time Frame: Baseline of PA0008, Week 48
Population: Subset of study participants in the FAS with Dactylitis at PA0008 Baseline (LDI>0).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Bimekizumab 160 mg (FAS)
Number analyzed (Participants) | 45
score on a scale | -54.31 (67.09)

9. Secondary Outcome: Percentage of Participants With Psoriasis Area Severity Index (PASI75) Response at Week 48 Calculated Relative to Baseline of PA0008
Description: The PASI75 response assessments are based on at least 75% improvement in the PASI score from Baseline of PA0008. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining percentage of skin covered with psoriasis (PSO) for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. For the Final score, minimum possible PASI value is 0= no disease, maximum value is 72= maximal disease. Missing PASI responses were imputed using least observation carried forward (LOCF) for any visits where the corresponding BSA has not increased compared to the preceding visit.
Time Frame: Baseline of PA0008, Week 48
Population: Subset of study participants in FAS with body surface area (BSA) affected by psoriasis of >=3% at PA0008 Baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 160 mg (FAS)
Number analyzed (Participants) | 120
percentage of participants | 90.0

10. Secondary Outcome: Percentage of Participants With Psoriasis Area Severity Index (PASI90) Response at Week 48 Calculated Relative to Baseline of PA0008
Description: The PASI90 response assessments are based on at least 90% improvement in the PASI score from Baseline of PA0008. Body divided into 4 areas: head, arms, trunk to groin, and legs to top of buttocks. Assignment of an average score for the redness, thickness, and scaling for each of the 4 body areas with a score of 0 (clear) to 4 (very marked). Determining percentage of skin covered with PSO for each of the body areas and converting to a 0 to 6 scale. Final PASI= average redness, thickness, and scaliness of the psoriatic skin lesions, multiplied by the involved psoriasis area score of the respective section, and weighted by the percentage of the person's affected skin for the respective section. For the final score, minimum possible PASI value is 0= no disease, maximum value is 72= maximal disease. Missing PASI responses were imputed using LOCF for any visits where the corresponding BSA has not increased compared to the preceding visit.
Time Frame: Baseline of PA0008, Week 48
Population: Subset of study participants in FAS with BSA affected by psoriasis of >=3% at PA0008 Baseline.
Measure: Number; unit: percentage of participants
Arm/Group | Bimekizumab 160 mg (FAS)
Number analyzed (Participants) | 120
percentage of participants | 80.0

ADVERSE EVENTS:
Time Frame: From Entry Visit of PA0009 until Safety Follow-Up Visit (up to Week 120)
Description: A TEAE was defined as an event with onset date on or after the start date of study medication in PA0009.
Arm/Group | Bimekizumab 160 mg (SS)
All-Cause Mortality (participants affected / at risk) | 0/183
Serious Adverse Events (participants affected / at risk) | 14/183
Other Adverse Events (participants affected / at risk) | 82/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bimekizumab 160 mg (SS) (N=183)
Anal fistula (Gastrointestinal disorders) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 2 (2)
Chronic sinusitis (Infections and infestations) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 2 (2)
Pregnancy on contraceptive (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 1 (1)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bimekizumab 160 mg (SS) (N=183)
Oral candidiasis (Infections and infestations) | 13 (23)
Bronchitis (Infections and infestations) | 11 (15)
Upper respiratory tract infection (Infections and infestations) | 20 (29)
Nasopharyngitis (Infections and infestations) | 19 (24)
Pharyngitis (Infections and infestations) | 10 (11)
Sinusitis (Infections and infestations) | 10 (10)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 12 (13)
Psoriasis (Skin and subcutaneous tissue disorders) | 14 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-12-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT03347110/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT03347110/SAP_001.pdf